CLINICAL TRIAL: NCT05868044
Title: REsponse to Combined SuPra-orbital and Occipital Nerve Stimulation in Chronic Cluster HeadachE with the PRIMUS System, a First in Human Study
Brief Title: REsponse to Combined SONS and ONS in Chronic Cluster HeadachE
Acronym: RESPONSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salvia BioElectronics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SCI-01-CCH
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRIMUS (Experimental): PRIMUS system
  Interventions: Device: PRIMUS

INTERVENTIONS:
Device: PRIMUS — PRIMUS system

SUMMARY:
The purpose of this study is to demonstrate the safe use of the PRIMUS System in subjects with chronic cluster headache. This is a single-centre, open label, prospective, first in human study to collect initial clinical data on the PRIMUS system for the treatment of chronic cluster headache.

ELIGIBILITY:
Main Inclusion Criteria:

* Able and willing to provide informed consent
* Documented chronic cluster headache for at least 1 year as per ICHD-3 criteria
* Attack frequency of ≥ 4 attacks per week for ≥ 4 weeks before enrolment
* Documented failure of verapamil (failure meaning ineffective, provoked unacceptable side-effects or contra-indicated)
* Stable on preventive treatment for at least two weeks prior to enrolment.
* Agree to refrain from starting new prophylactic cluster headache medication or other preventive treatments, from 4 weeks before entering the baseline period throughout the duration of the study
* MRI available (not older than 4 years prior to study enrolment) or willing to undergo an MRI to exclude structural lesions potentially causing headache
* Able and willing to complete a headache Diary

Main Exclusion Criteria:

* Any other chronic primary or secondary headache disorder, unless they can clearly differentiate them from cluster headache attacks based on the quality and associated symptoms
* Concomitant neuromodulation, except tVNS
* Previous failure to any implantable neuromodulation device for neurovascular headache
* Have an existing Active Implantable Medical Device nearby the implant location (e.g. DBS, cochlear implant, …)
* Metal implants in the skull (e.g. skull plates, seeds) nearby the implant
* Have a pacemaker or implantable cardioverter defibrillator (ICD)
* Suboccipital infiltrations with steroids and/or local anaesthetics or use of oral steroids in the past 3 months
* Use of botulinum toxin injections in the past 12 weeks
* Calcitonin gene-related peptide inhibitors started less than 12 weeks prior to enrolment
* Women of childbearing age who are pregnant, nursing or not using contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation | 4 weeks
  The primary safety assessment is the incidence of serious procedure and/or device-related adverse events in all subjects at 30 days.
Safety Evaluation | 12 months
  The primary safety assessment is the incidence of serious procedure and/or device-related adverse events in all subjects at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Frank, MD, Principal Investigator — Resolve Pain
Locations (1):
- Resolve Pain, Buderim, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No